CLINICAL TRIAL: NCT06118203
Title: Evaluation of Circulating Endothelial Inflammatory Biomarkers in Response to GLP-1 Agonist Semaglutide in Acute Pulmonary Embolism
Brief Title: Semaglutide Use in Acute Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 300440
Record Dates: First submitted 2023-09-11; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism | interventions — semaglutide

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Patient plasma samples, collected at baseline and at study completion 4 week time-point
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Open label Semaglutide: Patients presenting with acute intermediate - high risk PE consenting to participation in drug arm of study
  Interventions: Drug: Semaglutide
- Control: Patients presenting with acute intermediate - high risk PE consenting to participation in control arm of study

INTERVENTIONS:
Drug: Semaglutide — Semaglutide in addition to standard of care
  Other Names: None applicable
  Groups: Open label Semaglutide

SUMMARY:
Evaluation of circulating endothelial inflammatory biomarkers in response to GLP-1 agonist Semaglutide in acute pulmonary embolism

DETAILED DESCRIPTION:
Study Rationale and risk/benefit analysis

This GLP-1 intervention study in patients with acute PE represents an original hypothesis in a population with unmet clinical need. The results of this study could have important and immediate clinical implications in improving outcomes for this patient group. The current long-term treatment of acute PE is limited to anticoagulation, and there are no other studies investigating different treatment approaches. Vascular inflammation is known to be an important factor driving thrombus evolution and vascular remodelling, and therefore exploring the utility of targeting vascular inflammation is an important step forward in developing new treatment strategies for this common condition.

We aim to conduct a proof-of-concept open label study with biomarker response to evaluate Semaglutide, a GLP-1 agonist, administered as add-on therapy to the standard of care in adult patients with acute PE treated in hospital. Outcomes will be compared to a control group who will not receive the study drug. The study will recruit adult patients with proximal or large clot burden PE with evidence of right ventricular dysfunction on admission. This group has the highest risk of impaired clot resolution and of development of long-term complications including chronic thromboembolic disease.

There is a low risk of study drug complications given the extensive availability of human clinical trial data with GLP-1 agonists. There is also extensive real-world experience on the use of Semaglutide in the clinical investigation of glucose control in diabetes. As the first dose of the study drug is administered in hospital, clinical monitoring is optimised and common biochemical perturbations (hypoglycaemia) are easily interrogated and acted on by the clinical team. Patients who have contraindications to the use of GLP-1 agonists and patients currently taking GLP-1 agonists for diabetes mellitus are excluded to reduce the risks associated with the study drug even further.

Trial Objectives and Design

Trial Objectives

This proof-of-concept interventional study will comprise three separate but inter-linking aims:

I. Determine the effect of Semaglutide on highly glycosylated CD147- driven vascular inflammation in acute PE and GLP-1 receptor expression levels.

II. Evaluate immunological effects of Semaglutide in patients with acute PE (T cell receptor expression/cytokine, chemokine levels).

III. Determine the impact of Semaglutide on clot resolution and right ventricular recovery following acute PE.

4.2. Primary endpoints Evaluate the change in highly glycosylated CD147 between day 0 and following 6 weeks of Semaglutide.

4.3. Secondary endpoints I. Determine the rate of persistent CTPA or VQ scan perfusion defects with Semaglutide.

II. Change in right ventricular function, FAC andTASPE on echocardiography between day 0 and following 6 weeks of Semaglutide.

III. Change in plasma Cyclophylin A, sCD147, D-dimer, E selectin, VCAM, MMP levels, NTproBNP, GLP1-R, Troponin, myeloperoxidase activity.

ELIGIBILITY:
Inclusion Criteria:

Acute pulmonary embolism

Exclusion Criteria:

Concurrent use of GLP-1 agonist

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute admission with acute pulmonary embolism
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-03-04 (Actual); Study Completion 2023-03-05 (Actual)

PRIMARY OUTCOMES:
Endothelial biomarker measurement | 4 weeks
  Change in plasma CD147 level between baseline and 4 weeks

SECONDARY OUTCOMES:
Plasma proteomics | 4 weeks
  Change in plasma proteome between baseline and 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colm McCabe, MD, Principal Investigator — Imperial College London
Locations (1):
- Colm McCabe, London, United Kingdom

REFERENCES:
- [Derived] Samaranayake CB, Chen YC, Fang M, Rhodes CJ, Song S, Sabrin F, Ashek A, Bonnici K, Mukherjee B, Howard LS, Pinguel J, Rawal B, Semple T, Price LC, Wort SJ, Rudd T, Zhao L, McCabe C. GLP-1 agonist, semaglutide use in acute pulmonary embolism recovery: a four-week proof-of-concept study including proteomic profiling. Eur Heart J Open. 2025 Dec 24;6(1):oeaf170. doi: 10.1093/ehjopen/oeaf170. eCollection 2026 Jan. PMID 41536961